CLINICAL TRIAL: NCT00987961
Title: Linking Hospitalized Injection Drug Users to Buprenorphine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Michael Stein, MD, Principal Investigator, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA026223 (NIH)
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Opiate Dependence
Keywords: opioid dependence; suboxone; HIV risk behavior
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Genetic Linkage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as usual (No Intervention): Participants in this arm will receive the standard detox treatment for individuals hospitalized with opioid dependence.
- Linkage (Experimental): Participants in this arm will receive a maintenance schedule of Suboxone during their hospital stay, and an appointment with an outpatient Suboxone provider for after their discharge.
  Interventions: Behavioral: Linkage

INTERVENTIONS:
Behavioral: Linkage — This intervention provides an outpatient appointment with a Suboxone provider for medically hospitalized opioid-dependent patients to attend post-discharge.
  Arms: Linkage

SUMMARY:
This study tests whether starting Suboxone (buprenorphine) during a medical hospitalization, and then providing an appointment (a "link") for after discharge to maintenance buprenorphine in an outpatient setting will reduce HIV risk behavior in individuals who inject opioids.

DETAILED DESCRIPTION:
In this randomized controlled trial, medically hospitalized opioid dependent patients will be assigned to a "treatment as usual" group, where they will receive a detox regiment of Suboxone during their hospital stay, or a "linkage" group, where they receive a maintenance course of Suboxone during their hospital stay, and appointment post-discharge with an outpatient Suboxone clinic/provider and a Suboxone prescription to use between discharge and this appointment. Study interviews are completed at baseline, and 1, 3- and 6-months post-baseline. Primary outcomes are opioid use and HIV risk behavior.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Current opioid injector, at least weekly in the past month
* Current opioid dependence, SCID confirmed
* Currently receiving an inpatient buprenorphine detoxification protocol.

Exclusion Criteria:

* Patients unable to be interviewed due to acute illness or cognitive impairment
* In police custody, expecting incarceration
* Persons who cannot provide two contact persons (including shelters, parole officers, etc.) to verify location
* Not able to complete assessments in English
* Enrolled in a methadone maintenance program
* Plans to leave the area within the next 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2009-09; Primary Completion 2014-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
opioid use | baseline, 1-month, 3-months, 6-months
HIV risk behavior | baseline, 1-month, 3-months, 6-months

SECONDARY OUTCOMES:
reduction in injection-related medical conditions | baseline, 1-month, 3-months, 6-months
reduction in emergency department and hospital utilization | baseline, 1-month, 3-months, 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Stein, MD, Principal Investigator — Butler Hospital
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Liebschutz JM, Crooks D, Herman D, Anderson B, Tsui J, Meshesha LZ, Dossabhoy S, Stein M. Buprenorphine treatment for hospitalized, opioid-dependent patients: a randomized clinical trial. JAMA Intern Med. 2014 Aug;174(8):1369-76. doi: 10.1001/jamainternmed.2014.2556. PMID 25090173
- [Derived] Meshesha LZ, Tsui JI, Liebschutz JM, Crooks D, Anderson BJ, Herman DS, Stein MD. Days of heroin use predict poor self-reported health in hospitalized heroin users. Addict Behav. 2013 Dec;38(12):2884-7. doi: 10.1016/j.addbeh.2013.08.002. Epub 2013 Aug 14. PMID 24045030